CLINICAL TRIAL: NCT04093141
Title: Chemotherapy Followed by Irreversible Electroporation in Patients With Unresectable Locally Advanced Pancreatic Cancer (CHEMOFIRE-2)
Brief Title: Chemotherapy Followed by Irreversible Electroporation in Patients With Unresectable Locally Advanced Pancreatic Cancer
Acronym: CHEMOFIRE-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ole Thorlacius-Ussing, MD, DMSc, Professor of Surgery (Other)
Responsible Party: Sponsor-Investigator, Ole Thorlacius-Ussing, MD, DMSc, Professor of Surgery, Professor of surgery, Consultant surgeon, DMSc, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N-20190013
Record Dates: First submitted 2019-05-03; First posted 2019-09-17 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Unresectable Pancreatic Cancer
Keywords: locally advances pancreatic cancer; irreversible electroporation; nanoknife; phase II; efficacy
MeSH Terms: interventions — Electroporation

STUDY DESIGN:
Intervention Model Description: Patients in the study will be compared to data from clinical registry.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Intervention (Experimental)
  Interventions: Procedure: IRE

INTERVENTIONS:
Procedure: IRE — in situ irreversible electroporation
  Other Names: irreversible electroporation

SUMMARY:
This study is a single-arm clinical trial of irreversible electroporation (IRE) for the treatment of unresectable locally advanced pancreatic cancer (LAPC).

The aim of the study is to evaluate the efficacy of IRE in this patient group. A statistical analysis of patient survival will be performed, comparing study participants to historical data from the Danish national database of pancreatic cancer patients.

DETAILED DESCRIPTION:
Patients with unresectable LAPC can be included in the study. Prior to inclusion, initial treatment with chemotherapy with or without radiation therapy (RT) is administered to all patients accord to the referring institutions protocol. Some patients will have undergone an attempted resection prior to inclusion. It is expected, that a substantial number of patients are participants in the LAPC-03 protocol (FOLFIRINOX followed by local therapy (resection, RT and/or IRE) in patients with LAPC).

After completion of initial therapy, potential study participants are restaged with a PET-CT scan and serum tumor markers. Patients found on restaging to be free of metastatic disease and without significant primary tumor progression will be candidates for IRE therapy. IRE therapy will be administered not earlier than 2 weeks after completion of initial therapy.

IRE will be done under general anesthesia as an in-patient procedure. Patients will attend study specific visits with PET-CT scan 3, 6, 9, 12, 18 and 24 months post-IRE. Patients will attend the out-patient clinic after 1, 3, 6, 9, 12, 15, 18, 21 and 24 months. During this we will monitor pain, quality of life, global functioning and nutritional status.

In patients who, at any time during the study, are assessed as candidates for resection, a more detailed re-evaluation of resectability is performed according to local preferences (e.g. EUS and/or LAP/LUS and/or CT and/or MR).

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytologically proven adenocarcinoma/carcinoma of the pancreas.
* Largest tumor diameter ≤4 cm in any plane.
* >18 years of age.
* Prior treatment with neoadjuvant chemotherapy for at least 2 months
* Tumor must be deemed as unresectable at the national pancreatic multidisciplinary team conference after neoadjuvant treatment.
* Non-progressive disease according to Response Evaluation Criteria in Solid Tumors v1.1 (RECiST 1.1) after neoadjuvant treatment.
* Patients must be able to give informed consent.

Exclusion Criteria:

* Tumor is inaccessible e.g. due to venous dilation etc. (assessed with preoperative ultrasound).
* ASA score >3
* ECOG performance status >2
* Pregnancy.
* Atrial fibrillation.
* Implanted electronic device e.g. cardiac pacemakers or other electrostimulators.
* Metal stents or other metallic objects near the ablation zone (unless the stent can be replaced with a plastic stent prior to IRE).
* Signs of severe disease of the bone marrow, kidney or liver during time of treatment. Treatment may be postponed if the disease state is reversible.
* Severe allergies to anesthetic agent, paralytic agent or any of the equipment used during treatment.
* Patient is referred from hospital outside of Denmark

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
2-year survival proportion from 1) diagnosis and 2) IRE | 2 years after the last patient is enrolled

SECONDARY OUTCOMES:
Median overall survival from 1) diagnosis and 2) IRE | 2 years after the last patient is enrolled
Progression free survival after IRE | 2 years after the last patient is enrolled
Median time to local progression after IRE | 2 years after the last patient is enrolled
Median time to dissemination after IRE | 2 years after the last patient is enrolled
90-day complication rate and severity (Clavien-Dindo) | 90 days after the last patient is enrolled
Resection rate | 2 years after the last patient is enrolled
Quality of life (EORTC QLQ C-30) | Every 3 months for 2 years after the intervention
  Quality of life questionnaire - Core 30 is used to assess the quality of life in the included patients. Raw scores will be calculated according to the manual. Items will be grouped in: Global health status (range 0 - 100, high is good), Functional scales (range 0 - 100, high is good) and symptom scales (range 0 - 100 low is good). Differences in each scales during the course of the trial we be calculated seperately.
Perioperative pain perception (VAS) | Every week for 1 month after the intervention
  Perioperative pain will be scores using the visual analogue pain scale (range 0 - 10, low score is less pain).
Long term pain perception (m-BPI-SF) | Every 3 months for 2 years after the intervention
  Long term pain will be assessed using the modified Danish version of the Brief Pain Inventory - short form. The outcomes assessed will be an average score of pain severity items and interference items in accordance with the manual. The scales range from 0 to 10 (lower is less pain).
ECOG performance status | Every 3 months for 2 years after the intervention
  Physicians assessment of global functioning using the "Eastern Cooperative Oncology Group" perfomance status scale (range 0 - 5, low score is better)
Nutritional status assessment (PG-SGA-SF) | Every 3 months for 2 years after the intervention
  Nutritional status assessment using the Scored Patient-Generated Subjective Global Assessment (short form). The short form includes only patient reported measures and will be combined into a single score according to the manual (range 0 - 37,low score is better).

CONTACTS AND LOCATIONS:
Overall Officials: Ole Thorlacius-Ussing, Professor, DMSc, Principal Investigator — Department of gastrointestinal surgery, Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No